CLINICAL TRIAL: NCT05121363
Title: A Single-arm, Multicenter Phase II Clinical Trial to Evaluate TQB2858 Injection Combined With Anlotinib Hydrochloride Capsule in the Treatment of Recurrent or Metastatic Advanced Endometrial Cancer
Brief Title: A Clinical Trial to Evaluate TQB2858 Injection Combined With Anlotinib Hydrochloride Capsule in the Treatment of Recurrent or Metastatic Advanced Endometrial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2858-II-01
Record Dates: First submitted 2021-11-15; First posted 2021-11-16 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2858 injection + Anlotinib Hydrochloride capsules (Experimental): TQB2858 injection: once every 3 weeks, 1800mg each time, intravenous infusion. Until the disease progression or unbearable adverse events occur.
  Anlotinib Hydrochloride capsules: once a day,12mg each time, oral administration before breakfast. Continuous administration for 2 weeks, withdrawal for 1 week, i.e. 3 weeks (21 days) as a course of treatment. Until the disease progression or unbearable adverse events occur.
  Interventions: Drug: TQB2858 injection; Drug: Anlotinib Hydrochloride capsules

INTERVENTIONS:
Drug: TQB2858 injection — TQB2858 is an anti-programmed death receptor 1(anti-PD-1) /Transforming growth factor-β(TGF-β )bi-functional fusion protein
Drug: Anlotinib Hydrochloride capsules — Anlotinib Hydrochloride is a multi-target tyrosine kinase inhibitor.

SUMMARY:
A clinical trial to evaluate TQB2858 injection combined with Anlotinib Hydrochloride capsule in the treatment of recurrent or metastatic advanced endometrial carcinoma

ELIGIBILITY:
Inclusion Criteria:

Only those who meet all the following inclusion criteria can be enrolled in this study:

* (1) The subjects voluntarily joined the study, signed the informed consent form;
* (2) Age: 18 -75years old (when signing the informed consent); Performance status score: 0-1;The expected survival time is more than 3 months;
* (3) Endometrial carcinoma confirmed by histopathology;
* (4) Previous treatment with 1-2 line standard systemic chemotherapy regimen failed or intolerated;"intolerance" is defined as ≥ grade IV hematological toxicity or ≥ grade III non-hematological toxicity during treatment. Neoadjuvant or adjuvant chemotherapy is allowed in the early stage. If disease progression / recurrence occurs during neoadjuvant / adjuvant therapy or within 12 months after the end of treatment, neoadjuvant / adjuvant therapy is considered to be a first-line systemic chemotherapy failure for progressive diseases.
* (5)Confirmed to have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1.
* (6)The main organs function well and meet the following standards:

  1. Blood routine examination standards (correction without blood transfusion and hematopoietic stimulating factor drugs within 14 days before examination): Hemoglobin (HGB) ≥ 80 g / L；The absolute value of neutrophils (NEUT) ≥ 1.5x109 / L；Platelet count ((PLT)) ≥ 90 × 109 PG / L.
  2. Biochemical examination shall meet the following standards:Total bilirubin (TBIL) ≤ 1.5 times the normal upper limit (ULN);Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN. If with liver metastasis, ALT and AST ≤ 5 × ULN;Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance rate (Ccr) ≥ 60ml/min.
  3. Blood coagulation function should meet the following standards: international standardized ratio (INR) ≤ 1.5×ULN (no anticoagulant therapy or over five drug half-lives );
  4. Thyroid function examination should meet the following standards: the thyroid stimulating hormone (TSH) ≤ ULN; if abnormal, the levels of T3 and T4 should be examined. If the levels of T3 and T4 are normal, they can be selected.
  5. Evaluation by color Doppler echocardiography: left ventricular ejection fraction ((LVEF)) ≥ 50%
* (7) Female subjects of childbearing age should agree that contraceptive measures (such as IUDs or condoms) must be used during the study period and within 6 months after the end of the study; the serum pregnancy/urine pregnancy test is negative within 7 days before the study, and must be non-lactation subjects;male subjects should agree that contraceptive measures must be used during the study period and within 6 months after the end of the study

Exclusion Criteria:

Those who meet any of the following criteria will not be enrolled in this study:

* (1) Concomitant disease and medical history:

  1. Present or present with other malignant tumors within 2 years before medicine for the first time.The following two conditions can be included: other malignant tumors treated by single operation, disease-free survival (DFS) for 5 consecutive years; cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumor [Ta (non-invasive tumor), Tis (in situ) and T1 (tumor infiltrating basement membrane)]；
  2. Pathological diagnosis of uterine sarcoma, such as carcinosarcoma (malignant mullerian mixed tumor), endometrial leiomyosarcoma, endometrial stromal sarcoma or other high-grade sarcomas；
  3. There are a variety of factors that affect oral drugs (such as inability to swallow, chronic diarrhea and intestinal obstruction, etc.)
  4. Unalleviated toxicity higher than Common Terminology Criteria for Adverse Events (CTCAE) level 1 due to any previous antineoplastic therapy, excluding alopecia and peripheral sensory nerve disorders;
  5. Major surgical treatment or significant traumatic injury within 28 days prior to the start of study treatment (excluding needle aspiration, endoscopic biopsy for diagnostic purposes, etc.);
  6. A wound or fracture that has not been cured for a long time, possessing risk factors for fracture (such as bearing bone metastases, etc.)
  7. Within 6 months before initial administration, there have been arteriovenous thrombotic events such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism,etc;
  8. Those who have a history of psychotropic substance abuse and are unable to quit or have mental disorders;
  9. Subjects with any severe and / or uncontrolled disease,including:

     1. Blood pressure control is not satisfactory after standard treatment(systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 100mmHg).
     2. Patients who have experienced myocardial ischemia or myocardial infarction within six months; New York Heart Association(NYHA )grade ≥2 congestive heart failure; Grade ≥2 atrioventricular block; Arrhythmias that cannot be stably controlled with drugs (including corrected QT interva ≥470ms) and arrhythmias that may have a potential impact on trial treatment;
     3. Active infection ( CTCAE grade ≥ 2 infection);
     4. Decompensated liver cirrhosis, active hepatitis *;

        * active hepatitis (hepatitis B reference:Hepatitis B surface antigen( HBsAg )positive, and Hepatitis B virus DNA(HBV DNA)>2500 copies /mL or > 500 IU/mL; Hepatitis C reference: hepatitis C virus(HCV) antibody positive, and HCV virus titer test value exceeds the upper limit of normal value); Note: Subjects with positive surface antigen of hepatitis B or positive core antibody and hepatitis C patients eligible for inclusion are advised to continue antiviral therapy to prevent virus activation;
     5. Active syphilis and active tuberculosis;
     6. Renal failure requiring hemodialysis or peritoneal dialysis: glomerular filtration rate(eGFR) < 15ml/ (min•1.73㎡);
     7. A history of immunodeficiency, including Human Immunodeficiency Virus( HIV) positive or other acquired or congenital immunodeficiency disease, or a history of organ transplantation;
     8. Poor control of diabetes (Fasting blood glucose (FBG) > 10mmol/L, bedtime blood glucose > 11.1mmol/L and hemoglobin A1C (HbA1c) ≥8.5% before bedtime);
     9. Patients with urine protein ≥++ as indicated by routine urine examination, and 24-hour urine protein quantity > 1.0g;
     10. Persons suffering from epilepsy and requiring medical treatment.
* (2) Tumor-related symptoms and treatment:

  1. Received surgery, chemotherapy, radiation or other anticancer therapy within 4 weeks before the start of study treatment (the wash out period is calculated from the end of the last treatment); Those who had previously received local radiation therapy were eligible to enroll if they met the following criteria: the end of radiotherapy was more than 4 weeks before the start of study therapy (brain radiation was more than 2 weeks); The target lesions selected in this study are not in the radiotherapy region; or the target lesion is located in the radiotherapy area, but progression is confirmed.
  2. Received the treatment of Chinese patent medicines with anti-tumor indications specified in the National Medical Products Administration(NMPA) approved drug instructions (including compound cantharidin capsules, Kangai injection, Kanglaite capsule/injection, Aidi injection, brucea javanica oil injection/capsule, Xiaoaiping tablet/injection, Huachansu capsule, etc.) within 2 weeks before the study treatment;
  3. Previously received immunomodulator therapy, including therapeutic vaccines, cytokine therapy, or Anti-programmed death receptor 1(anti-PD-1), Programmed death ligand-1(PD-L1), Cytotoxic T lymphocyte-associated protein 4(CTLA-4), High purity recombinant protein（4-1BB）, T cell activation markers（OX-40） and other related immunotherapy drugs;
  4. Previous use of anti-angiogenic drugs such as bevacizumab, anlotinib, apatinib, lenvatinib, sorafenib, sunitinib, regorafenib, fruquintinib, etc.(applicable to the stage 2; stage 1: not include bevacizumab;
  5. Received hormone therapy for endometrial cancer within 1 week prior to the first dose of trial drug (for endometrioid cancer only)
  6. Pleural effusion, pericardial effusion, or ascites that uncontrolled and still requires repeated drainage (as determined by the investigator);
  7. Imaging (CT or MRI) showed that the tumor had invaded the important blood vessels or was judged by the researchers to be most likely to invade the important blood vessels and cause fatal massive hemorrhage during the follow-up study.
  8. Subjects with known central nervous system metastasis and / or cancerous meningitis; unless asymptomatic or treated and stable, no imaging evidence of new brain metastasis or enlarged brain metastasis was found at least 4 weeks after brain metastasis treatment, and steroid or anticonvulsant therapy was stopped for at least 14 days before the start of the study.
* (3) Research treatment related:

  1. Have a history of live attenuated vaccine administration within 28 days before the start of study treatment or planned live attenuated vaccine administration during the study period;
  2. Have a history of severe allergy to Anlotinib Hydrochloride capsule or known components of TQB2858 injection;
  3. An active autoimmune disease requiring systemic treatment (such as palliative drugs, corticosteroids, or immunosuppressants) occurred within 2 years before the start of study therapy. Alternative therapies (such as thyroxine, insulin, or physical corticosteroids for adrenal or pituitary dysfunction, etc.) are not considered systemic treatment;
  4. Diagnosed as immunodeficient or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose >10mg/ d of prednisone or other equivalent hormone) and continued use within 2 weeks of initial administration;
* (4) Participated in clinical trials of other antitumor drugs within 4 weeks before initial administration or no exceeding drug' 5 half-lives.
* (5)According to the researcher's judgment, subjects who have concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or who are considered unsuitable for inclusion for other reasons.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Baseline up to two years
  Proportion of patients whose tumors shrank by a certain amount and remained for a certain period of time, including complete response (CR) and partial response (PR) cases

SECONDARY OUTCOMES:
Progress Free Survival (PFS) | Baseline up to two years
  The period from the first use of the drug to disease progression or death (whichever occurs first)
Disease Control Rate (DCR) | Baseline up to two years
  Proportion of subjects whose tumors shrink or remain stable for a certain period, including complete remission（CR）, partial remission（PR） and stable disease（SD）;
Duration of Response (DOR) | Baseline up to two years
  The period from firstly-recorded objective tumor response (CR or PR) to firstly-recorded objective tumor progression or death due to any cause (whichever occurs first) .
Overall Survival (OS) | Baseline up to two years
  The period from the first use of the drug to death from all causes. For subjects who are still alive at the last follow-up, the OS will be counted as data censored based on the last follow-up. For subjects who are lost follow-up, the OS will be counted as data censored based on the last confirmed survival time before being lost to follow-up.
Incidence of adverse events: Occurrence of all adverse events (AE), serious adverse events (SAE), and treatment-related adverse events (TEAEs) | Baseline up to two years
  AEs refer to all adverse medical events that occur after a patient or clinical trial subject receives an experimental drug, which can be expressed as symptoms, signs, diseases, or abnormalities in laboratory tests, but are not necessarily related to the treatment of the experimental drug. SAEs refer to adverse medical conditions such as death, life threatening, permanent or severe disability, loss of function, the need for hospitalization or prolonged hospitalization , and congenital abnormalities or birth defects after the subject receives the experimental drug

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hunan Cancer Hospita, Changsha, Hunan
  - Qilu Hospital of Shandong University, Jinan, Shandong